CLINICAL TRIAL: NCT06924970
Title: A Phase 2, Double-blind, Randomized, Placebo-Controlled, Multicenter, Dose- Finding, Efficacy, and Safety Study of Tebapivat in Participants With Sickle Cell Disease
Brief Title: A Dose-Finding Study of Tebapivat to Assess Efficacy, and Safety in Participants With Sickle Cell Disease (SCD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG946-C-003; 2024-519746-70-01 (EU CTIS Number)
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tebapivat 2.5 milligrams (mg) (Experimental): Participants will receive 2.5 mg tebapivat orally, once daily (QD) for 12-weeks in the double-blind (DB) period. Participants who complete the DB Period will be eligible to receive the same dose in the Open-Label Extension (OLE) period for up to 52 weeks.
  Interventions: Drug: Tebapivat
- Tebapivat 5.0 mg (Experimental): Participants will receive 5.0 mg tebapivat orally, QD, for 12-weeks in the DB period. Participants who complete the DB Period will be eligible to receive the same dose in the OLE period for up to 52 weeks.
  Interventions: Drug: Tebapivat
- Tebapivat 7.5 mg (Experimental): Participants will receive 7.5 mg tebapivat orally, QD, for 12-weeks in the DB period. Participants who complete the DB Period will be eligible to receive the same dose in the OLE period for up to 52 weeks.
  Interventions: Drug: Tebapivat
- Tebapivat Matched Placebo (Placebo Comparator): Participants will receive a matched placebo, orally, QD, for 12-weeks in the DB period. Participants who complete the DB Period will be randomized in 1:1:1 to receive tebapivat 2.5 mg QD, tebapivat 5.0 mg QD, or tebapivat 7.5 mg QD in the OLE period for up to 52 weeks
  Interventions: Drug: Tebapivat; Drug: Tebapivat Matched Placebo

INTERVENTIONS:
Drug: Tebapivat — Oral tablets.
  Other Names: AG-946
Drug: Tebapivat Matched Placebo — Oral tablets.
  Arms: Tebapivat Matched Placebo

SUMMARY:
The main purpose of this study is to compare the effect of tebapivat versus placebo on anemia and to detect a dose-response for hemoglobin (Hb) response in participants with SCD.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of SCD (HbSS, HbSC [combined heterozygosity for hemoglobins S and C], sickle hemoglobin [HbS]/β0-thalassemia, HbS/β+-thalassemia, or other sickle cell syndrome variants).
* Hemoglobin ≥5.5 and ≤10.5 grams per decilitre (g/dL). Hemoglobin concentration must be based on an average of at least 2 Hb concentration measurements (separated by ≥7 days) collected during the screening period.
* If taking hydroxyurea, the hydroxyurea dose must be stable for at least 90 days before randomization. Discontinuation of hydroxyurea requires a 90-day washout before providing informed consent.

Key Exclusion Criteria:

* Receiving regularly scheduled red blood cell (RBC) transfusion therapy (also termed chronic, prophylactic, or preventative transfusion); episodic transfusion in response to worsened anemia or vaso-occlusive crisis (VOC) is permitted. Additionally, a participant who requires episodic transfusion(s) may not have received a transfusion(s) within 60 days before providing informed consent or during the screening period.
* >10 sickle cell pain crisis (SCPCs) in the 12 months before providing informed consent.
* Receiving anabolic steroids that have not been stopped for at least 4 weeks before randomization. Testosterone replacement therapy to treat hypogonadism is allowed; the testosterone dose and preparation must be stable for ≥10 weeks before randomization.
* Hospitalized for an SCPC and/or other vaso-occlusive event within 14 days before providing informed consent or within 14 days before randomization. If an SCPC occurs during the screening period, the screening period may be extended with Medical Monitor approval.
* Receiving treatment with voxelotor, crizanlizumab, or L-glutamine within 90 days before randomization.
* Platelet count <lower limit of normal (LLN) for the local laboratory or <150×109/liter (L) (whichever is lower) during screening. Platelet transfusions received within 28 days before consent or during screening.
* Receiving treatment with hematopoietic stimulating agents within 90 days before randomization.
* Prior exposure to gene therapy or prior bone marrow or stem cell transplantation, including any conditioning regimen.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Hb Response | Baseline, Week 10 through Week 12

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 72
Average Change From Baseline in Hb Concentration | Baseline, Week 10 through Week 12
Average Change From Baseline in Indirect Bilirubin | Baseline, Week 10 through Week 12
Average Change From Baseline in Lactate Dehydrogenase (LDH) | Baseline, Week 10 through Week 12
Average Change From Baseline in Absolute Reticulocyte Count | Baseline, Week 10 through Week 12
Average Change From Baseline in Percent Reticulocytes | Baseline, Week 10 through Week 12
Average Change From Baseline in Erythropoietin | Baseline, Week 10 through Week 12
Average Change From Baseline in Patient Reported Outcomes Measurement Information System® (PROMIS) Fatigue 13a Short Form Score | Baseline, Week 10 through Week 12
Average Change From Baseline in PROMIS Pain Intensity 1a Score | Baseline, Week 10 through Week 12
Average Change From Baseline in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Impact Score | Baseline, Week 10 through Week 12
Plasma Concentration of Tebapivat | Pre-dose and at multiple timepoints post-dose up to Week 8
Maximum (Peak) Concentration (Cmax) of Tebapivat | Pre-dose and at multiple timepoints post-dose up to Week 8
Time to Cmax (tmax) of Tebapivat | Pre-dose and at multiple timepoints post-dose up to Week 8
Area Under the Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-t) of Tebapivat | Pre-dose and at multiple timepoints post-dose up to Week 8
Whole Blood Concentrations of 2,3-Diphosphoglycerate (2,3-DPG) | Pre-dose and at multiple timepoints post-dose up to Week 8
Whole Blood Concentrations of Adenosine Triphosphate (ATP) | Pre-dose and at multiple timepoints post-dose up to Week 8

CONTACTS AND LOCATIONS:
Locations (31):
- United States (16):
  - UCHealth at University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UConn Health, Farmington, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Medical Center & Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lifespan at Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Farris Road, Greenville, South Carolina
  - University of Texas Health Science Center of Houston, Houston, Texas
  - Fred Hutchinson Cancer Center, University of Washington, Seattle, Washington
- Belgium (2):
  - CHR de la Citadelle, Liège, Wallonne
  - Clinique CHC MontLégia, Liège, Wallonne
- Canada (3):
  - Scarborough Health Network - Centenary Hospital, Scarborough Village, Ontario
  - CHU Montreal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- France (3):
  - Hôpital Edouard Herriot, CHU de Lyon, Lyon, Auvergne-Rhône-Alpes
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, Midi Pyrenees
  - CHU Hôpital Henri Mondor, Créteil, Île-de-France Region
- St. James Hospital, Dublin, Leinster, Ireland
- Netherlands (3):
  - Amsterdam Universitair Medisch Centrum, Locatie AMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- United Kingdom (3):
  - Evelina London Children's Hospital, Guy's and St. Thomas' NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No